CLINICAL TRIAL: NCT05160194
Title: Gaining Real-Life Skills Over the Web (GROW)
Brief Title: Gaining Real-Life Skills Over the Web
Acronym: GROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90IFDV0003
Record Dates: First submitted 2021-08-30; First posted 2021-12-16 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Parent-Child Relations; Parenting
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GROW Intervention (Other): Every participant received the GROW Intervention, chose not to participate in the GROW intervention, or dropped out before completing the GROW Intervention.
  Interventions: Behavioral: Positive Parenting Intervention

INTERVENTIONS:
Behavioral: Positive Parenting Intervention — The highly interactive GROW Program consists of 5 core modules and 1 optional, supplemental session. Each session is expected to take 15-20 minutes to complete, and at the end of each module, parents record a 5 minute "special play time" video interacting with their child to demonstrate the skills they learned in the session. Each online module is followed by a meeting with a trained therapist who will discuss their "special play time" video and the skills they are learning. Parents make their way through the 5 core modules sequentially before accessing the supplemental session that may be relevant to them.

SUMMARY:
Gaining Real-life Skills Over the Web (GROW) is an online parenting-skills intervention for caregivers of children aged 0-4 who sustained traumatic brain injuries. GROW is designed to promote family and child coping and adjustment for caregivers.

DETAILED DESCRIPTION:
This project develops and evaluates an online learning environment of web-based intervention modules designed to promote family and child coping and adjustment (GROW: Gaining Real-life Skills Over the Web) based on a comprehensive needs assessment of children aged 0 to 14 years old, who experienced a traumatic brain injury (TBI) between the ages of 0 to 4 years, and their families. The incidence of TBI peaks between the ages 0 to 4 years, yet there are no evidenced-based interventions to facilitate neurocognitive development and socio-emotional functioning of children injured during this critical development period. To address the unmet need of caregivers of infants and toddlers with TBI, the project uses a three-phase development process to generate proof of concept and initial proof of product. Phase 1 involves a comprehensive needs assessment that includes quantitative assessment of family and child needs, qualitative assessment through focus groups and interviews of families, feedback from family and professional advisory boards, and consultation with professionals implementing interventions with similar populations (e.g., families of children with very low birth weight). During Phase 2, the project develops the content and manual for the intervention modules, designs the online learning environment, and conducts intensive, iterative usability testing. Phase 3 involves a pilot of the GROW program with 20 families to evaluate its usability, acceptability, and qualitative and quantitative impact on stakeholder identified outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age at injury and enrollment: ages 0-4, inclusive
2. Overnight hospitalization for traumatic brain injury
3. Mechanism of injury: Non-penetrating traumatic brain injury; abusive head trauma (AHT) will be included
4. Language: English must be the primary spoken language in the home

Exclusion Criteria:

1. Does not reside with the caregiver at least half-time
2. The caregiving situation is not stable (i.e., there must be no scheduled custody hearings)
3. English is not the primary language spoken in the home
4. Families of children who are non-responsive or in a persistent vegetative state will also be excluded
5. Caregivers with a psychiatric hospitalization in the past year will be ineligible to participate
6. If AHT is the suspected injury mechanism, the child must not reside with the suspected abuser, must have been in the current living situation for at least 6 months, and must be anticipated to remain in this living situation for the next 6 months. The study team will only recruit non-abusing caregivers (including foster parents) to participate.

Ages: 0 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression(CES-D) Scale Change | Pre-Intervention and Immediately Post-Intervention
  Measuring caregiver psychological distress, the CES-D consists of 20 items that are rated on a 4-point likert scale (from 1: rarely or none of the time to 4: most or all of the time). Scores range from zero to sixty. Higher scores indicated a higher frequency of depressive symptoms during the last week.
Parenting Stress Index (PSI) Change | Pre-Intervention and Immediately Post-Intervention
  The study team used the 36 item short form PSI to measure caregiver stress. Using a 4-point likert scale, the stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Patient-Reported Outcomes Measurement Information System Change | Pre-Intervention and Immediately Post-Intervention
  The study team used only the Sleep, Stress, and Anxiety Measures which are rated on a 5-point likert scale. Each measure has a range in score from 7 to 35 with higher scores indicating greater severity.
Family Burden of Injury Interview (FBII) Change | Pre-Intervention and Immediately Post-Intervention
  The FBII measures family burden. Open-ended answers are coded Yes/No and are given a stress rating of 0 (not at all)-5(extremely stressful). Caregiver responses are averaged to provide an index of injury-related family burden.
MacArthur-Bates Communicative Development Inventories (MB-CDI) Change | Pre-Intervention and Immediately Post-Intervention
  Using the short form MB-CDIs to measure child language abilities, the scoring scale is a minimum of 0- maximum of 310 with greater scores showing better language abilities.
Caregiver-Child Observation Change | Pre-Intervention and Immediately Post-Intervention
  Using the Parent/Child Toy Play Ratings in the Play and Learning Strategies (PALS) manual, 6 domains (warmth, contingent responsiveness, demonstration/physical teaching, verbal stimulation/scaffolds, restrictions, and negativity/intrusiveness) are rated on scales of 1 to 5 with 1 being the worst rating and 5 being the best.
GROW Satisfaction Survey | Immediately Post-Intervention
  Satisfaction with intervention measured in both 5-point likert scale ratings (with higher values showing greater satisfaction) and open-ended feedback about participant experience in the program.
Background & Family Information Form | Pre-Intervention
  Demographics rehabilitation services

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Maggard BL, Gies LM, Sidol CA, Moscato EL, Schmidt M, Landry SH, Makoroff KL, Rhine TD, Wade SL. Online Intervention for Caregivers of Children with Early Traumatic Brain Injury: Pilot Trial. J Pediatr Psychol. 2023 Mar 20;48(3):205-215. doi: 10.1093/jpepsy/jsac080. PMID 36240452